CLINICAL TRIAL: NCT02529189
Title: A Randomised, Double-blind, Placebo-controlled Study Investigating the Effects of Dietary Nitrate on Vascular Function, Platelet Reactivity and Restenosis in Stable Angina
Brief Title: Investigating the Effects of Dietary Nitrate on Vascular Function, Platelet Reactivity and Restenosis in Stable Angina
Acronym: NITRATE-OCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/LO/0555
Record Dates: First submitted 2015-08-07; First posted 2015-08-20 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Stable Angina; Angioplasty; Optical Coherence Tomography; Nitrate
MeSH Terms: conditions — Cardiovascular Diseases; Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): 70 ml of a beetroot juice concentrate containing ~5 mmol nitrate
  Interventions: Dietary Supplement: Beetroot Juice
- Nitrate-deplete beetroot juice (Placebo Comparator): 70 ml of a beetroot juice concentrate that is nitrate-depleted
  Interventions: Dietary Supplement: Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — 70 ml of beetroot juice containing ~5 mmol of inorganic nitrate
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Beetroot Juice — 70 ml of beetroot juice which is nitrate-depleted
  Arms: Nitrate-deplete beetroot juice

SUMMARY:
The mainstay treatment for reducing the symptoms of angina and long-term risk of heart attacks in patients with heart disease is stent implantation in the diseased coronary artery. Whilst this procedure has revolutionised treatment the incidence of secondary events remains a concern. These repeat events are due in part to continued enhanced platelet reactivity, endothelial dysfunction and a phenomenon called 'restenosis' i.e. the stent becomes blocked ultimately requiring another expensive and risky procedure. In this study it will be determined whether a once daily inorganic nitrate administration might favourably modulate platelet reactivity and endothelial function leading to a decrease in restenosis.

DETAILED DESCRIPTION:
To address the aims a proof-of-concept study will be conducted to ascertain whether a dietary nitrate approach might prove useful adjunctive therapy improving vascular function in patients with stable angina post elective angioplasty.

Design: A prospective randomised, single-centre, double-blind, placebo-controlled trial

Setting: Patients with stable angina and single/multiple coronary artery stenosis undergoing elective percutaneous coronary intervention (PCI) who are haemodynamically stable (systolic BP>100 mmHg). These patients will be recruited at The Barts Health Heart Centre, based at St. Bartholomew's Hospital. This is one of the biggest centres in the United Kingdom, serving a population of almost two million people from The City of London and The North East up to the M25 and is a 24/7 centre performing approximately 2000 non-primary angioplasties a year.

The study will take place in the Clinical Trials Unit, William Harvey Heart Centre.

Target population: A total of 300 patients (male and female, age 18-85) with stable angina as per requirements indicated above. Follow-up will take place in the Clinical Trials Unit, William Harvey Research Institute.

Treatment: Patients will be randomised (using an on line randomisation database) to receive 70 ml of a beetroot juice concentrate containing 4-5 mmol nitrate or nitrate-deplete placebo juice concentrate. This intervention will be taken by the patient daily from one day prior to re-establishment of flow with PCI and stent implantation.

Analysis: We will analyse the results based on an intention to treat analysis. We will also carry out further per protocol analyses and a subgroup analysis on patients who are on organic nitrates as part of their routine therapy and a comparison of DES (drug-eluting stents) versus BMS (bare-metal stents).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable angina diagnosed by a cardiologist on optimal medical therapy undergoing angioplasty to treat residual symptoms.
2. Aged 18-85
3. Patients able and willing to give their written informed consent.
4. Patients undergoing successful PCI procedure.

Exclusion Criteria:

1. Unstable ischaemic heart disease, with an episode of chest pain in less than 24 hours.
2. Patients who have had previous coronary artery bypass surgery (CABG), if they are undergoing angioplasty within a non-native vessel.
3. Patients undergoing angioplasty with a bio-absorbable stent.
4. Current diagnosis of or treatment for malignancy, other than non-melanoma skin cancer.
5. Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
6. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
7. Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
8. Severe acute infection, or significant trauma (burns, fractures).
9. Pregnancy. This will be tested by urine human chorionic gonadotropin (hCG) measurement
10. History of alcohol or drug abuse within the past 6 months.
11. A history of heart failure New York Heart Association (NYHA) class 3-4 or severe left ventricular dysfunction (left ventricular ejection fraction of <30%) regardless of symptom status.
12. Systemic autoimmune disease such as rheumatoid arthritis, connective tissue disease, or other conditions known to be associated with chronic inflammation such as inflammatory bowel disease.
13. Patients who have donated > 500mls blood within 56 days prior to study medication administration.
14. Anaemia with Hb <10g/dl, or any other known blood disorder or significant illness that may affect platelet function, and coagulation.
15. A history of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody or other chronic hepatic disorder) or HIV.
16. Abnormal liver function due to acute or chronic liver conditions 3 x upper limit of normal at screening.
17. Renal impairment with creatinine clearance (eGFR) of 35ml/min at screening.
18. If patients are on mouthwash, they must be willing to stop using this at least 1 week before the start of the study and throughout the duration that they are involved in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Difference between groups in In-stent late loss, where late loss is defined as the difference between the minimum luminal diameter (MLD). | 6 months +/- 1 month post intervention

SECONDARY OUTCOMES:
Difference from baseline within the group and between groups in endothelial function assessed by flow-mediated dilatation of the brachial artery at 6 months compared to pre-procedure assessment. | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in target vessel revascularisation (TVR). | 6 months post intervention
Difference from baseline within the group and between groups in restenosis rate (diameter >50%). | 6 months post intervention
Difference from baseline within the group and between groups in in-segment late loss. | 6 months post intervention
Difference from baseline between groups in major adverse cardiac events (i.e. Myocardial Infarction, death, Cerebrovascular Accident, Target Vascular Revascularisation). | 6 months, 12 months and 24 months post intervention
Difference from baseline within the group and between groups in inflammatory markers. | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in plasma and erythrocyte nitrite reductase. | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in changes in plasma xanthine oxidase activity. | 6 months and 12 months post intervention
Difference from baseline within the group and between groups high-sensitivity C-reactive protein (hsCRP). | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in Interleukin-6 (IL-6). | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in platelet activation (P-Selectin and platelet-monocyte aggregates). | 6 months and 12 months post intervention
Difference from baseline within the group and between groups in platelet aggregation ex vivo (ADP, collagen, arachidonic acid). | 6 months and 12 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- William Harvey Research Institute, Barts and The London School of Medicine, London, United Kingdom

REFERENCES:
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Ghosh SM, Kapil V, Fuentes-Calvo I, Bubb KJ, Pearl V, Milsom AB, Khambata R, Maleki-Toyserkani S, Yousuf M, Benjamin N, Webb AJ, Caulfield MJ, Hobbs AJ, Ahluwalia A. Enhanced vasodilator activity of nitrite in hypertension: critical role for erythrocytic xanthine oxidoreductase and translational potential. Hypertension. 2013 May;61(5):1091-102. doi: 10.1161/HYPERTENSIONAHA.111.00933. Epub 2013 Apr 15. PMID 23589565
- [Derived] Rathod KS, Mathur A, Shabbir A, Khambata RS, Lau C, Beirne AM, Chhetri I, Ono M, Belgaid DR, Massimo G, Ramasamy A, Tufaro V, Jain AK, Poulter N, Falaschetti E, Jones DA, Garcia-Garcia HM, Bourantas C, Learoyd A, Warren HR, Ahluwalia A. The NITRATE-OCT study-inorganic nitrate reduces in-stent restenosis in patients with stable coronary artery disease: a double-blind, randomised controlled trial. EClinicalMedicine. 2024 Oct 18;77:102885. doi: 10.1016/j.eclinm.2024.102885. eCollection 2024 Nov. PMID 39469537
- [Derived] Rathod KS, Jones DA, Van-Eijl TJ, Tsang H, Warren H, Hamshere SM, Kapil V, Jain AK, Deaner A, Poulter N, Caulfield MJ, Mathur A, Ahluwalia A. Randomised, double-blind, placebo-controlled study investigating the effects of inorganic nitrate on vascular function, platelet reactivity and restenosis in stable angina: protocol of the NITRATE-OCT study. BMJ Open. 2016 Dec 20;6(12):e012728. doi: 10.1136/bmjopen-2016-012728. PMID 27998900